CLINICAL TRIAL: NCT05439343
Title: Comparison of Analgesic Efficacy and Functional Improvement of Adductor Canal Block and Multimodal Local Infiltration Analgesia for Patients After Bilateral Total Knee Arthroplasty
Brief Title: Adductor Canal Block and Multimodal Local Infiltration Analgesia in Patients Receiving Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TPEVGH IRB No.: 2016-04-010C
Record Dates: First submitted 2022-05-19; First posted 2022-06-30 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Arthroplasty, Replacement, Knee; Analgesia; Rehabilitation
Keywords: Arthroplasty, Replacement, Knee; adductor canal block; Local infiltration; Regional analgesia; Pain, Postoperative; Rehabilitation; Muscle power
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Motion

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-centered, double-blinded, randomized controlled trial. We intend to compare two methods of postoperative analgesia, adductor canal block (ACB) and multimodal local infiltration (LI), simultaneously in patients receiving bilateral total knee arthroplasty. In other words, the patient will receive ACB in one knee and LI in the other knee after TKA surgery. Because this study is designed to apply these two methods respectively on either knee of the same patient, the relative analgesic efficacy can be assessed simultaneously. Like matched-pair designed study, this method can eliminate some confounding factors affecting pain scores.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor will not know which kind of interventions (adductor canal block and local infiltration) is performed on which knee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Experimental): Allocation of which limb is to receive adductor canal block is determined by randomization, using a computer-generated random sequence and opaque sealed envelopes. After completion of the TKA surgery and surgical suturing, adductor canal block will be performed by an anesthesiologist. Under ultrasound guidance, the femoral artery and the saphenous nerve are identified in the middle one-third of the thigh, deep to the sartorious muscle in the adductor canal. The sartorious and adductor muscles form the roof and the floor of the canal, respectively. Following skin infiltration, 20 mL of 0.25% bupivacaine with 1:400000 epinephrine is injected through a 3-inch, 23-gauge, short bevel block needle.
  Interventions: Other: Pain scores (numerical rating scale at rest and motion); Other: Secondary outcomes
- Local infiltration (Experimental): Allocation of the other limb to receive local infiltration is determined after randomization of the knee allocated for adductor canal block in the same patient. The chosen knee is infiltrated by the orthopedic surgeon intraoperatively with a 150-ml mixture of 150 mg bupivacaine, 10 mg morphine, 30 mg ketorolac, and 0.5 mg epinephrine. The posterior capsule is infiltrated before placement of the prosthesis, and the periarticular and superficial soft tissues are infiltrated after the prosthesis is in place and before wound closure.
  Interventions: Other: Pain scores (numerical rating scale at rest and motion); Other: Secondary outcomes

INTERVENTIONS:
Other: Pain scores (numerical rating scale at rest and motion) — As the primary outcome of the present clinical study, pain scores will be assessed with numerical rating scale at both rest and motion on both knees.
Other: Secondary outcomes — Brief Pain Inventory (Short Form), WOMAC Osteoarthritis index, and Lower extremity functional scale will be used as the questionnaires for functional assessment. Rehabilitation physiotherapy will be assessed with knee range of motion (both active and maximal passive), muscle power at abduction and adduction, single leg stance test, six-minute walk test for assessment of the functional recovery of knee joints.

SUMMARY:
Total knee arthroplasty (TKA) is associated with moderate to severe pain after operation. There are twenty thousand patients undertaking TKA annually in Taiwan, and the average length of hospital stay is about seven to ten days. In contrast, the length of hospital stay is only three to six days in some literatures. Adequate pain relief after surgery allows patients to mobilize earlier and easier and rehabilitate to reduce the length of hospital stay. By reducing hospital stay, we can reduce medical expenditure of national health insurance. In addition, effective analgesia can reduce the occurrence of chronic post-surgical pain which would compromise life quality and produce socioeconomic problems. This study tries to find a better solution for postoperative analgesia of TKA for patients in Taiwan. The present clinical study compares the effect of adductor canal block and local infiltration on postoperative analgesia and functional activity after TKA. To assess the outcome of both methods in the same patient, we can have more comparative result of pain score and functional parameters like range of motion of knee joint, time and ability to ambulate. Based on that, we try to find a better option for postoperative analgesia for patients receiving TKA in Taiwan.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with moderate to severe pain after operation. There are twenty thousand patients undertaking TKA annually in Taiwan, and the average length of hospital stay is about seven to ten days. In contrast, the length of hospital stay is only three to six days in some literature. Some patients choose to receive bilateral TKA simultaneously to avoid repetitive surgery and anesthesia, and are supposed to suffer more than those receiving unilateral TKA. Adequate pain relief after surgery allows patients to mobilize earlier and easier and rehabilitate to reduce the length of hospital stay and postoperative complications. By reducing the length of in-hospital stay and post-operative complication, we can reduce medical expenditure of national health insurance. In addition, effective analgesia can reduce the occurrence of chronic post-surgical pain which would compromise life quality and produce socioeconomic problems. This study tries to find a better solution for postoperative analgesia of TKA for patients in Taiwan. The present clinical study compares the effect of adductor canal block and local infiltration on postoperative analgesia and functional activity after bilateral simultaneous TKA. To assess the outcome of both methods in the same patient, we can have more comparative result of pain score and functional parameters like range of motion of knee joint, muscle power in knee adduction/abduction movement, and time and ability to ambulate. Based on that, we try to find a better option for postoperative analgesia for patients receiving TKA in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible to enter the study if their age are between 20 to 90 years old and scheduled for bilateral TKA secondary to osteoarthritis.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class IV-V, history of abnormal liver enzymes, hepatic failure, renal insufficiency, cardiac failure, organ transplant, neuropathic pain, history of stroke or major neurological deficit, coagulopathy, thrombocytopenia, sensory and motor disorders in lower limb, previous drug dependency, chronic use of opioids, allergy to local anesthetics and drug used in experiment, inability to walk independently, inability to comprehend pain assessment and patients refusing to have spinal anesthesia or enter this study.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | Baseline (the day before surgery)
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 2 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 8 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 24 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 36 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 48 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 60 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Hour 72 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | The day of discharge
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,
Pain score | Month 3 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable,

SECONDARY OUTCOMES:
Knee range of motion | Baseline (the day before surgery)
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Knee range of motion | Hour 24 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Knee range of motion | Hour 72 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Knee range of motion | the day of discharge
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Knee range of motion | Month 3 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Knee muscle power | Baseline (the day before surgery)
  Both adduction and abduction muscle power on both knees will be assessed with Commander Echo Algometry (pounds)
Knee muscle power | Hour 24 after surgery
  Both adduction and abduction muscle power on both knees will be assessed with Commander Echo Algometry (pounds)
Knee muscle power | Hour 72 after surgery
  Both adduction and abduction muscle power on both knees will be assessed with Commander Echo Algometry (pounds)
Knee muscle power | the day of discharge
  Both adduction and abduction muscle power on both knees will be assessed with Commander Echo Algometry (pounds)
Knee muscle power | Month 3 after surgery
  Both adduction and abduction muscle power on both knees will be assessed with Commander Echo Algometry (pounds)
Six minute walk test | Baseline (the day before surgery)
  To assess the walk ability (6-minute walk distance) before and after TKA surgery (meters)
Six minute walk test | Hour 24 after surgery
  To assess the walk ability (6-minute walk distance) before and after TKA surgery (meters)
Six minute walk test | Hour 72 after surgery
  To assess the walk ability (6-minute walk distance) before and after TKA surgery (meters)
Six minute walk test | the day of discharge
  To assess the walk ability (6-minute walk distance) before and after TKA surgery (meters)
Six minute walk test | Month 3 after surgery
  To assess the walk ability (6-minute walk distance) before and after TKA surgery (meters)
Single leg stance test | Baseline (the day before surgery)
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Single leg stance test | Hour 24 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Single leg stance test | Hour 72 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Single leg stance test | the day of discharge
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Single leg stance test | Month 3 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Functional questionnaires | Baseline (the day before surgery)
  Functional pain scale will be assessed with Western Ontario and McMaster Universities Osteoarthritis Index, Brief pain inventory (BPI) short form, and Lower extremity functional scale
Functional questionnaires | the day of discharge
  Functional pain scale will be assessed with Western Ontario and McMaster Universities Osteoarthritis Index, Brief pain inventory (BPI) short form, and Lower extremity functional scale
Functional questionnaires | Month 3 after surgery
  Functional pain scale will be assessed with Western Ontario and McMaster Universities Osteoarthritis Index, Brief pain inventory (BPI) short form, and Lower extremity functional scale
Adverse events | Baseline (the day before surgery)
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 2 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 8 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 24 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 36 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 48 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 60 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 72 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | the day of discharge
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Month 3 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia

CONTACTS AND LOCATIONS:
Overall Officials: Hsu Ma, MD, PhD, Study Chair — Institutional Review Board, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No